CLINICAL TRIAL: NCT01505491
Title: Pharmacokinetics and Safety of BI 695501 in Healthy Subjects: a Randomized, Open-label, Single Dose, Parallel Arm, Active Comparator Clinical Phase I Study
Brief Title: Pharmacokinetics and Safety Study of BI 695501 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1297.1
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2018-10

CONDITIONS: Healthy
MeSH Terms: interventions — Adalimumab

ARMS (3):
- BI 695501 (Experimental): Subject to receive one subcutaneous (s.c.) injection from a prefilled syringe containing BI 695501
  Interventions: Drug: BI695501
- adalimumab - US (Active Comparator): Subject to receive one s.c. injection from a prefilled syringe containing 40mg adalimumab
  Interventions: Drug: adalimumab
- adalimumab - EU (Active Comparator): Subject to receive one s.c. injection from a prefilled syringe containing 40mg adalimumab
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — 40mg adalimumab single s.c. injection
  Arms: adalimumab - EU
Drug: BI695501 — BI 695501 single s.c injection
  Arms: BI 695501
Drug: adalimumab — 40mg adalimumab single s.c. injection
  Arms: adalimumab - US

SUMMARY:
This trial will investigate the pharmacokinetics, safety and tolerability of BI 695501 and to establish pharmacokinetic equivalence of BI 695501 to adalimumab.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males
2. Body mass index (BMI) =18.5 to =29.9 kg/m2

Exclusion criteria:

1. Any clinically relevant abnormal finding of the medical examination (including blood pressure, pulse rate and electrocardiogram) deviating from normal and of clinical relevance
2. Any evidence of a clinically relevant previous or concomitant disease as judged by the investigator.
3. Chronic or relevant acute infections. A negative result for Human Immunodeficiency Virus, Hepatitis B and Hepatitis C testing is required for participation.
4. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
5. Intake of prescribed or over-the-counter drugs with a long half-life (>24 hours) within at least one month or less than 5 half-lives of the respective drug prior to administration or during the trial
6. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
7. Inability to refrain from smoking during days of confinement at the study center
8. Alcohol abuse (average more than 30 g/day)
9. Current drug abuse

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 193 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2012-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- New Zealand (2):
  - 1297.1.002 Boehringer Ingelheim Investigational Site, Auckland
  - 1297.1.001 Boehringer Ingelheim Investigational Site, Christchurch

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was phase I, open-label, randomised, parallel-arm, single-dose, active -comparator study with healthy subjects.
Pre-assignment Details: Subjects were screened for eligibility to participate in the trial. They attended a specialist sites which ensured strict implementation of inclusion/exclusion criteria and they were not to be entered in trial if any one of the specific entry criteria was violated. They were free to withdraw their consent at any time without penalty or prejudice.
Groups:
- BI 695501: Subject received one subcutaneous injection via prefilled syringe containing 40 milligram (mg) /0.8 milliliter (mL) BI 695501
- Humira®US: Subject received one subcutaneous injection via prefilled syringe containing 40 milligram (mg) /0.8 milliliter (mL) Humira®US
- Humira®EU: Subject received one subcutaneous injection via prefilled syringe containing 40 milligram (mg) /0.8 milliliter (mL) Humira®EU
Period: Overall Study
Arm/Group | BI 695501 | Humira®US | Humira®EU
Started | 67 | 62 | 64
Completed | 65 | 61 | 59
Not Completed | 2 | 1 | 5
Not completed — Other reason not listed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This set included all entered subjects who were treated with study medication and were documented to have received one dose of study drug. The TS contained all 193 subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 695501 | Humira®US | Humira®EU | Total
Number analyzed (Participants) | 67 | 62 | 64 | 193
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated Set
  Years | 26.3 (8.2) | 24.4 (6.6) | 27.6 (8.9) | 26.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    Female | 0 | 0 | 0 | 0
    Male | 67 | 62 | 64 | 193
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was not captured in this trial Population: Treated Set
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 10 | 7 | 7 | 24
    Native Hawaiian or Other Pacific Islander | 1 | 3 | 1 | 5
    Black or African American | 0 | 1 | 1 | 2
    White | 56 | 51 | 55 | 162
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the BI 695501 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the BI 695501 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞). Geometric mean and geometric coefficient of variation (gCV) are provided as descriptive statistic.
Time Frame: 1 hour (h) before drug administration and 1, 4, 8, 12, 24, 48, 60, 72, 84, 96, 108, 120, 132, 144, 168, 192, 240, 312, 480, 648, 816, 1032, 1320, 1704 h after drug administration
Population: Pharmacokinetic set (PKS): This set included all subjects of the randomized and treated set who in addition provided at least one Pharmacokinetic (PK) endpoint and had no important protocol violations relevant to the evaluation of bio-equivalence.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micro-gram*hour/milliliter (μg*h/mL)
Arm/Group | BI 695501 | Humira®US | Humira®EU
Number analyzed (Participants) | 67 | 62 | 64
Micro-gram*hour/milliliter (μg*h/mL) | 2740 (48.2) | 2390 (44.3) | 2050 (53.2)
Statistical Analysis 1: Comparison: BI 695501 vs Humira®US; ANOVA (analysis of variance) model on the logarithm scale was used with 'treatment' and 'age' as fixed effect; Test type: Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.1163, ANOVA; Geometric mean ratio (%) = 113.22, 90% CI 2-sided [98.752 to 129.812], Standard Error of Mean 1.086 — Bio-equivalence of BI 695501 vs. Humira US was estimated by the ratios of the adjusted geometric means (gMean). Standard error of the mean is actually geometric standard error
Statistical Analysis 2: Comparison: BI 695501 vs Humira®EU; ANOVA (analysis of variance) model on the logarithm scale was used with 'treatment' and 'age' as fixed effect; Test type: Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.7345, ANOVA; Geometric mean ratio (%) = 132.24, 90% CI 2-sided [113.984 to 153.412], Standard Error of Mean 1.094 — Bio-equivalence of BI 695501 vs. Humira EU was estimated by the ratios of the adjusted geometric means (gMean). Standard error of the mean is actually geometric standard error
Statistical Analysis 3: Comparison: Humira®US vs Humira®EU; ANOVA (analysis of variance) model on the logarithm scale was used with 'treatment' and 'age' as fixed effect; Test type: Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.1833, ANOVA; Geometric mean ratio (%) = 86.51, 90% CI 2-sided [74.974 to 99.830], Standard Error of Mean 1.090 — Bio-equivalence of Humira EU vs. Humira US was estimated by the ratios of the adjusted geometric means (gMean). Standard error of the mean is actually geometric standard error

2. Primary Outcome: Area Under the Concentration-time Curve of the BI 695501 in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the BI 695501 in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz). Geometric mean and geometric coefficient of variation (gCV) are provided as descriptive statistic.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micro-gram*hour/milliliter (μg*h/mL)
Arm/Group | BI 695501 | Humira®US | Humira®EU
Number analyzed (Participants) | 67 | 62 | 64
Micro-gram*hour/milliliter (μg*h/mL) | 2480 (40.0) | 2250 (37.7) | 1890 (46.1)
Statistical Analysis 1: Comparison: BI 695501 vs Humira®US; ANOVA (analysis of variance) model on the logarithm scale was used with 'treatment' and 'age' as fixed effect; Test type: Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.0303, ANOVA; Geometric mean ratio (%) = 109.42, 90% CI 2-sided [97.384 to 122.935], Standard Error of Mean 1.073 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 695501 vs Humira®EU; ANOVA (analysis of variance) model on the logarithm scale was used with 'treatment' and 'age' as fixed effect; Test type: Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.6547, ANOVA; Geometric mean ratio (%) = 128.88, 90% CI 2-sided [113.492 to 146.365], Standard Error of Mean 1.080 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Humira®US vs Humira®EU; ANOVA (analysis of variance) model on the logarithm scale was used with 'treatment' and 'age' as fixed effect; Test type: Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.1572, ANOVA; Geometric mean ratio (%) = 86.24, 90% CI 2-sided [76.238 to 97.564], Standard Error of Mean 1.077 — [estimate comment as in outcome 1, analysis 3]

3. Primary Outcome: Maximum Measured Concentration of the BI 695501 in Plasma (Cmax)
Description: Maximum measured concentration of the BI 695501 in plasma (Cmax). Geometric mean and geometric coefficient of variation (gCV) are provided as descriptive statistic.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micro-gram/milliliter (μg/mL)
Arm/Group | BI 695501 | Humira®US | Humira®EU
Number analyzed (Participants) | 67 | 62 | 64
Micro-gram/milliliter (μg/mL) | 4.47 (34.2) | 4.07 (34.2) | 3.74 (40.5)
Statistical Analysis 1: Comparison: BI 695501 vs Humira®US; ANOVA (analysis of variance) model on the logarithm scale was used with 'treatment' and 'age' as fixed effect; Test type: Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.0212, ANOVA; Geometric mean ratio (%) = 110.30, 90% CI 2-sided [99.687 to 122.035], Standard Error of Mean 1.063 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 695501 vs Humira®EU; ANOVA (analysis of variance) model on the logarithm scale was used with 'treatment' and 'age' as fixed effect; Test type: Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.1700, ANOVA; Geometric mean ratio (%) = 117.53, 90% CI 2-sided [105.638 to 130.757], Standard Error of Mean 1.066 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Humira®US vs Humira®EU; ANOVA (analysis of variance) model on the logarithm scale was used with 'treatment' and 'age' as fixed effect; Test type: Equivalence — p-value for ratio outside interval 80% to 125%; p = 0.0016, ANOVA; Geometric mean ratio (%) = 96.53, 90% CI 2-sided [87.064 to 107.017], Standard Error of Mean 1.064 — [estimate comment as in outcome 1, analysis 3]

4. Secondary Outcome: Terminal Half- Life of the BI 695501 in Plasma (t1/2)
Description: Terminal half- life of the BI 695501 in plasma (t1/2).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | BI 695501 | Humira®US | Humira®EU
Number analyzed (Participants) | 67 | 62 | 64
hour | 292 (104) | 230 (76.8) | 236 (98.3)

5. Secondary Outcome: Apparent Clearance of the BI 695501 in the Plasma After Extra-vascular Administration (CL/F)
Description: Apparent clearance of the BI 695501 in the plasma after extra-vascular administration (CL/F).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per minute (mL/min)
Arm/Group | BI 695501 | Humira®US | Humira®EU
Number analyzed (Participants) | 67 | 62 | 64
Milliliter per minute (mL/min) | 0.244 (48.2) | 0.279 (44.3) | 0.326 (53.2)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until end of the study, up to 79 days
Arm/Group | BI 695501 | Humira®US | Humira®EU
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/62 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/62 | 0/64
Other Adverse Events (participants affected / at risk) | 35/67 | 29/62 | 33/64
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 (N=67) | Humira®US (N=62) | Humira®EU (N=64)
Upper respiratory tract infection (Infections and infestations) | 13 | 10 | 17
Rhinitis (Infections and infestations) | 5 | 1 | 1
Headache (Nervous system disorders) | 17 | 16 | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 1
Fatigue (General disorders) | 4 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.